CLINICAL TRIAL: NCT05359926
Title: Early Versus Delayed Urinary Catheter Removal After Minimally Invasive Lumbar Spine Surgery: A Randomized-Controlled Clinical Trial
Brief Title: Early Versus Delayed Urinary Catheter Removal After Minimally Invasive Lumbar Spine Surgery
Acronym: EDUCaRe
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Benefits of no foley outweighed enrollment and use of foley.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Brandon Carlson, MD, MPH, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00148694
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-10

CONDITIONS: Foley Catheterization; Ambulation
Keywords: lumbar spine; foley catheterization; ambulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Urethral Catheter Removal (Experimental): Removal of the urethral catheter in the operating room at the conclusion of surgery
  Interventions: Other: Experimental
- Delayed Urethral Catheter Removal (Active Comparator): Removal of the urethral catheter in next morning after surgery
  Interventions: Other: Active comparator

INTERVENTIONS:
Other: Experimental — Early urethral foley removal after the surgery
  Arms: Early Urethral Catheter Removal
Other: Active comparator — Delayed urethral foley removal after the surgery
  Arms: Delayed Urethral Catheter Removal

SUMMARY:
The study aims to compare between early versus delayed urinary catheter removal the impact on time to ambulation (in minutes) after minimally invasive lumbar spine surgery

DETAILED DESCRIPTION:
Early ambulation enables rapid removal of drainage tubes and canisters and decreases length of hospitalization. Previous article showed that a 1-day shorter in hospitalization led to an approximately US$ 2000 reduction in total patient costs. Another study examining patients after total knee arthroplasty found that an early discharge group, a decrease in length of stay in 22h resulted in financial savings of approximately US$ 600 per case.

Another author found that early ambulation was associated with 19% lower 90-day readmission rate. Moreover, early ambulation contributed to 50.6% lower probability of developing at least one complication than regular ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Minimally invasive one- or two-level lumbar fusion procedures

Exclusion Criteria:

* Patients that cannot give consent
* Patients with lower extremity amputation(s);
* Non-minimally invasive surgeries
* Patients with pre-existing bladder/kidney or urinary tract dysfunction
* Patients with spinal cord injuries
* Patients with known lower extremity weakness and impaired mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Ambulation | After the surgery, postoperative day 1
  Time in minutes to ambulation

SECONDARY OUTCOMES:
Facility discharge | Average postoperative day 1-3
  Number of subjects discharge to facility
Home discharge | Average postoperative day 1-3
  Number of subjects discharge to home
Hospital length of stay | 1 to 3 days
  Total number of days in the hospital
Pain medication | Hospitalization period: postoperative day 1, 2, 3
  Total dose of opioid medication in milligrams used by each subject
Urinary catheter reinsertion | From date of the surgery until the date of first documented event, whichever came first, assessed up to discharge (1 to 3 days) after the surgery
  Total number of urinary catheter reinsertion
Urinary tract infection | From date of the surgery until the date of first documented event, whichever came first, assessed up to 1 month after the surgery
  Total number of urinary tract infection after urinary catheter removal
Physical therapy progression | Hospitalization period: postoperative day 1, 2, 3
  Maximum walking distance tolerated in meters by each subject

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Carlson, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang J, Shi Z, Duan FF, Fan MX, Yan S, Wei Y, Han B, Lu XM, Tian W. Benefits of Early Ambulation in Elderly Patients Undergoing Lumbar Decompression and Fusion Surgery: A Prospective Cohort Study. Orthop Surg. 2021 Jun;13(4):1319-1326. doi: 10.1111/os.12953. Epub 2021 May 7. PMID 33960687
- [Background] Gornitzky AL, Flynn JM, Muhly WT, Sankar WN. A Rapid Recovery Pathway for Adolescent Idiopathic Scoliosis That Improves Pain Control and Reduces Time to Inpatient Recovery After Posterior Spinal Fusion. Spine Deform. 2016 Jul;4(4):288-295. doi: 10.1016/j.jspd.2016.01.001. Epub 2016 Jun 16. PMID 27927519
- [Background] Raudenbush BL, Gurd DP, Goodwin RC, Kuivila TE, Ballock RT. Cost analysis of adolescent idiopathic scoliosis surgery: early discharge decreases hospital costs much less than intraoperative variables under the control of the surgeon. J Spine Surg. 2017 Mar;3(1):50-57. doi: 10.21037/jss.2017.03.11. PMID 28435918
- [Background] Marsh J, Somerville L, Howard JL, Lanting BA. Significant cost savings and similar patient outcomes associated with early discharge following total knee arthroplasty. Can J Surg. 2019 Feb 1;62(1):20-24. doi: 10.1503/cjs.002118. PMID 30265646
- [Background] Park P, Nerenz DR, Aleem IS, Schultz LR, Bazydlo M, Xiao S, Zakaria HM, Schwalb JM, Abdulhak MM, Oppenlander ME, Chang VW. Risk Factors Associated With 90-Day Readmissions After Degenerative Lumbar Fusion: An Examination of the Michigan Spine Surgery Improvement Collaborative (MSSIC) Registry. Neurosurgery. 2019 Sep 1;85(3):402-408. doi: 10.1093/neuros/nyy358. PMID 30113686